CLINICAL TRIAL: NCT03798405
Title: Reactive vs. Proactive Pain Control in Hospitalized Patients With Inflammatory Bowel Disease
Brief Title: Reactive vs. Proactive Pain Control in IBD
Acronym: PAIN-Sparing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19-related restrictions
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Gil Melmed, co-Director, Inflammatory Bowel Disease Center, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Pro00050742
Record Dates: First submitted 2018-12-04; First posted 2019-01-10 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Inflammatory Bowel Diseases; Pain; Opioid Use; Crohn Disease; Ulcerative Colitis
Keywords: Pain; Inflammatory Bowel Disease; Opioids
MeSH Terms: conditions — Inflammatory Bowel Diseases; Pain; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Consecutive patients with IBD admitted to the hospital will be screened, and eligible patients will be consented. Patients who have a pain score > 0 and require pain control will randomly receive the reactive traditional prescribing or the proactive standard-of-care orderset guideline - all patients will receive a FitBit exercise tracker.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary investigators will be blinded, as will the computer programmers who collect the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive (Experimental): Proactive Analgesic Inpatient Narcotic-Sparing:
  Pain management in patients in the proactive physician-behavior group will be based on the IBD Pain orderset in our EMR. This orderset is already in use and standard-of-care at Cedars. The orderset uses pain medications, which have evidence for use in IBD. The orderset is simply a guide to clinicians and does not force any doctor or patient to be in a "protocol".
  Interventions: Behavioral: Proactive Analgesic Inpatient Narcotic-Sparing
- Reactive (Control Group) (No Intervention): Pain management in patients in the reactive group (control group) will follow traditional prescribing habits. As different providers vary in the way they treat pain, analgesic medication prescribing in the control group will be inherently variable in nature. The control group does not constitute a lack of treatment or placebo; rather, pain management in the control group will not be proactive as in the intervention group.

INTERVENTIONS:
Behavioral: Proactive Analgesic Inpatient Narcotic-Sparing — Medications suggested to the physician with enhanced ease of ordering.
  Other Names: P.A.I.N.-Sparing Bundle
  Arms: Proactive

SUMMARY:
The investigators will compare two physician behaviors for managing pain in patients with IBD: proactive vs. reactive. Both the proactive and reactive behavior/strategies are standard of care at the institution in which the study will be performed. The PROACTIVE strategy is an IBD-specific analgesic orderset (built into our EMR and approved by the institution's Pharmacy and Therapeutics committee), the REACTIVE strategy is a traditional "reactive" analgesic prescribing (prescribing medications only when patients have pain). The PROACTIVE IBD-specific analgesic orderset consists of medications which have evidence for use in IBD-related pain. This orderset is an educational guide, it does not force any order. The reactive prescribing habits could contain an array of pain medications depending on what the provider wants to prescribe.

Aims:

Aim 1: To assess whether there is a difference in pain scores or functional activity among hospitalized patients with IBD between reactive vs proactive physician behaviors.

Aim 2: To assess whether there is a difference in inpatient opioid-prescribing between reactive vs proactive physician behaviors.

Aim 3: To assess whether there is a difference in health care utilization, including length-of-stay and 30-day readmission, between reactive vs proactive physician behaviors.

DETAILED DESCRIPTION:
Prospective, investigator-blinded, single-institution randomized-control trial . Consecutive adult patients with IBD (Crohn's disease or ulcerative colitis) admitted to the hospital will be screened for eligibility, and eligible patients will be approached and consented to participate. Subjects will be randomized to receive the P.A.I.N.-Sparing bundle or usual care. Patient randomization will be stratified by provider to avoid bias, using a web-based in-house system (RANDI3). Subjects will also be provided with a fitness tracker (Fitbit(R)) to measure functional status during their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Adults with confirmed IBD diagnosis
* Admitted for primary IBD-related sign or symptom

Exclusion Criteria:

* Admitted for primary non-IBD complaint
* Surgery in the last 30 days
* Alternative (non-IBD) GI diagnosis determined
* Age <18
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Pain Scores | Difference in the average daily pain score from the first to the last day of hospitalization, typically 7 days.
  Visual Analog Pain Numeric Rating Scale (Scale range 0 (no pain) to 10 (severe pain))

SECONDARY OUTCOMES:
Healthcare Utilization | From hospital admission until hospital discharge, typically 7 days.
  Hospital length of stay (in days)
Functional Activity | From hospital admission until hospital discharge, typically 7 days.
  FitBit activity (number of steps per day)
Opioid-Consumption | From hospital admission until hospital discharge, typically 7 days.
  Milligram morphine-equivalents consumed per day

CONTACTS AND LOCATIONS:
Overall Officials: Gil Y Melmed, MD, MS, Principal Investigator — Cedars-Sinai Medical Center; Sameer K Berry, MD, MBA, Study Director — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry SK, Takakura W, Patel D, Govalan R, Ghafari A, Kiefer E, Huang SC, Bresee C, Nuckols TK, Melmed GY. A randomized controlled trial of a proactive analgesic protocol demonstrates reduced opioid use among hospitalized adults with inflammatory bowel disease. Sci Rep. 2023 Dec 16;13(1):22396. doi: 10.1038/s41598-023-48126-0. PMID 38104145